CLINICAL TRIAL: NCT00285402
Title: Intranasal AST-726 Treatment for Prophylaxis of Migraine: A Placebo-Controlled Clinical Study
Brief Title: Efficacy and Safety Clinical Trial of Intranasal AST-726 for the Prevention of Migraine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ariston Pharmaceuticals, Inc. (Industry)
Responsible Party: John A. McLane, Ariston Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARPH-Cl-03; Eudract no: 2005-003349-15
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Migraine; Migraine Headache; Migraine Disorders; Migraine With Aura; Migraine Without Aura
Keywords: Migraine; Migraine prophylaxis; Migraine prevention; Chronic migraine treatment
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: AST-726 Low dose
- B (Experimental)
  Interventions: Drug: AST-726 High dose
- C (Placebo Comparator)
  Interventions: Drug: AST-726 Placebo

INTERVENTIONS:
Drug: AST-726 Low dose
  Arms: A
Drug: AST-726 High dose
  Arms: B
Drug: AST-726 Placebo
  Arms: C

SUMMARY:
The purpose of this migraine prevention study is to evaluate the efficacy and safety of AST-726 in moderate to severe migraine patients at one of two doses compared to placebo and compared to a baseline period as measured by a reduction in the number of migraine days.

DETAILED DESCRIPTION:
Migraine patients may experience repeated migraine attacks, lasting from four hours to three days or more. Each attack is characterized by severe pain, typically on one side of the head and often involves a number of other symptoms, including pain with a pulsating or throbbing quality, nausea or vomiting, sensitivity to light and sound, visual disturbances or aura. Currently the management of migraine may be either acute treatment or prophylaxis. Acute migraine treatment aims at aborting or reversing already present migraine symptoms with acute administration of medicine such as with triptans, whereas migraine prophylaxis aims to reduce the frequency and severity of migraine attacks over time through chronic medication.

The overall protocol design and outcome measurements of this study follow the guidelines and durations recommended by the International Headache Society for prophylaxis studies of migraine medications.

The study ARPH-CL-03 is a multicenter, randomized, double-blind, three parallel group design with moderate to severe migraine patients to assess the ability of daily administration of AST-726 at one of two doses to reduce the number of headache days in a 4 week period more than in patients that receive a placebo. AST-726 and the placebo will be self-administered by intranasal spray daily for 12 weeks. Among other efficacy and safety assessments, patients will have be asked to collect information on a daily migraine diary.

Patients will be instructed on the allowed use of acute migraine medications during this study.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Has migraine headaches with or without aura according to International Headache Society guidelines (Committee, 2004).
2. Has had migraines for at least 6 months prior to study enrollment period.
3. Migraines began before age 50.
4. Has 2 to 10 attacks per month and greater than or equal to 3 migraine days per month in the last 3 months prior to study enrollment.
5. Has 2 to 10 attacks in 30 days during the Baseline Period.

Additional inclusion criteria in protocol

Primary Exclusion Criteria:

1. Has headache equal to or greater than 18 days per month.
2. Has used migraine medications (e.g., topiramate, beta-blockers) for prophylactic use within 60 days prior to study enrollment.
3. Has excessive use of acute migraine medications (e.g., triptans, dihydroergotamine [DHE]) greater than 15 days per month.
4. Has taken nitroglycerine-containing medications within 60 days prior to study enrollment.
5. Failed more than 3 clinical studies of effective migraine prevention medications due to uncontrolled migraines.

Additional exclusion criteria in protocol

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable will be change in number of migraine headache days during standardized 30-day observation periods during treatment period and baseline period. The number of headache days reported in the patient diary will be standardized. | 30 days

SECONDARY OUTCOMES:
1 Number of subjects that respond with at least a 50% decrease in migraine days in each given 4-week Treatment Period | 4 weeks
2 The number of migraine headache attacks in each treatment period | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: W. M. Mulleners, Principal Investigator — Canisius-Wilhelmina Zeikenhuis
Locations (19):
- Finland (5):
  - Mediwest Research Centre Oy, Koskenalantie 16, Seinajoki
  - Turun Headache Center, Ltd. (Turun Paansarkykeskus Oy), Brahenkatu 11D, Turku, Turku
  - Suomen Terveystalo Jyvaskyla, Jyväskylä, Vainonkatu 30
  - Headache Center, Tammertutka, Hameenkatu 18 6th Floor, Tampere
  - Porin Laakerikeskus, Itsenalsyydenk. 33, Pori
- Netherlands (4):
  - Isala Kliniek, Groot Wezenland 20, Zwolle
  - Ziekenhuisgroep Twente, Afdeling Neurolgie , Locatie Streekziekenhuis Midden Twente, Geerdinksweg 141, Hengelo
  - St Anna Hospital, Bogardeind 2, Geldrop
  - Canisius Wilhelmina Hospital, Afdeling C02.04, Weg Door Jonkerbos 100 SZ Nimegen
- United Kingdom (10):
  - The Fowey River Practice; Rawlings Lane, Fowey, Cornwall
  - The Alverton Practice, 7 Alverton Terrace, Penzance, Cornwall
  - Saltash Health Centre, Saltash, Cornwall
  - The Staploe Medical Centre, Soham, Eky
  - Stonehill Medical Centre, Piggot st., Farnworth BL4 9QZ Bolton, Lancashire
  - Stanwell Road Surgery, 25 Stanwell Road, Ashford, Middlesex
  - The Circle Practice/Belmont Health Centre, Harrow, Middlesex
  - Woolwell Medical Centre, Devon, Plymouth
  - The Medical Centre, Kingston ave, East Horsley, Surrey
  - Albany House Medical Centre, 3 Queen St., Wellingborough